CLINICAL TRIAL: NCT04259788
Title: An AHEI Dietary Intervention to Reduce Pain in Women With Endometriosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Holly Harris, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RG1004314; 8772 (Other: FHCRC IRB Number); R01NR017951 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-02-06 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis
Keywords: Diet
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive in-person dietary counseling from a registered dietitian to help participants consume a diet that is consistent the AHEI dietary guidelines. Participants in this arm will be asked to consume this diet for a 12-week period and discontinue any vitamin or supplement intake during this time. During the first 4 weeks 2 meals and 1 snack/day will be shipped to the participant. During the last 8 weeks of the intervention, the study will provide the participants with a 14-day meal plan (3 meals and 2 snacks) that adheres to the AHEI maximum score criteria to help facilitate adherence to the diet.
  Interventions: Other: AHEI diet
- Control (No Intervention): Participants in this arm will not receive the dietary intervention.

INTERVENTIONS:
Other: AHEI diet — Main intervention is the consumption of an AHEI diet for 12 weeks.
  Arms: Intervention

SUMMARY:
The investigators are conducting this study to examine if a healthy diet based on the Alternative Healthy Eating Index (AHEI) influences pain symptoms, quality of life, and inflammatory markers measured in blood samples in women with endometriosis who are currently experiencing pain symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-45
* Laparoscopically-confirmed endometriosis
* Premenopausal (at least one period in the past 6 months)
* VAS pain score of at least 7 out of 10 in the previous 3 months
* Score below 75 on the AHEI-2010

Exclusion Criteria:

* Postmenopausal
* Pregnant
* Have had a hysterectomy or oophorectomy
* Have chronic illnesses that are known to affect gastrointestinal absorption of nutrients (celiac disease, Crohn's disease, ulcerative colitis, or cystic fibrosis)
* A history of kidney stones, cancer (except basal cell carcinoma), or diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain Measurement | Baseline
  Pain will be measured with components of the EPHect participant questionnaire using the VAS pain score. Scores range from 0 to 10, higher score is more pain (worse).
Pain Measurement | Baseline
  Pain will be measured with components of the EPHect participant questionnaire using the pain catastrophizing scale. Scores range from 0 to 52, higher scores indicate a greater amount of catastrophizing (worse).
Pain Measurement | Baseline
  Pain will be measured with components of the EPHect participant questionnaire using the mean number of analgesic and/or opioid pills taken per week.
Quality of Life Questionnaire | Baseline
  Physical and mental QOL components will be measured with the Endometriosis Health Profile Questionnaire. Scores range from 0 to 100, higher scores reflect more symptoms and worse health status.
Quality of Life Survey | Baseline
  Physical and mental QOL components will be measured with the Short Form-12 survey. There are two components, a physical component summary (PCS) and a mental health component summary (MCS). Both have a range of 0 to 100, higher scores represent better health.
Inflammatory Markers | Baseline
  Measurement of circulating levels of inflammatory markers (interleukin (IL)-6 and IL-1β.
Protein Measurement | Baseline
  Measurement of circulating levels of high sensitivity-C-reactive protein.
Tumor Necrosis Factor Measurement | Baseline
  Measurement of circulating levels of soluble tumor necrosis factor (TNF) alpha-receptor 1.
Tumor Necrosis Factor Measurement #2 | Baseline
  Measurement of circulating levels of soluble TNF alpha-receptor 2.
Pain Measurement | Week 4
  Pain will be measured with components of the EPHect participant questionnaire using the VAS pain score. Scores range from 0 to 10, higher score is more pain (worse).
Pain Measurement | Week 4
  Pain will be measured with components of the EPHect participant questionnaire using the pain catastrophizing scale. Scores range from 0 to 52, higher scores indicate a greater amount of catastrophizing (worse).
Pain Measurement | Week 4
  Pain will be measured with components of the EPHect participant questionnaire using the mean number of analgesic and/or opioid pills taken per week.
Quality of Life Questionnaire | Week 4
  Physical and mental QOL components will be measured with the Endometriosis Health Profile Questionnaire. Scores range from 0 to 100, higher scores reflect more symptoms and worse health status.
Quality of Life Survey | Week 4
  Physical and mental QOL components will be measured with the Short Form-12 survey. There are two components, a physical component summary (PCS) and a mental health component summary (MCS). Both have a range of 0 to 100, higher scores represent better health.
Inflammatory Markers | Week 4
  Measurement of circulating levels of inflammatory markers (interleukin (IL)-6 and IL-1β.
Protein Measurement | Week 4
  Measurement of circulating levels of high sensitivity-C-reactive protein.
Tumor Necrosis Factor Measurement | Week 4
  Measurement of circulating levels of soluble tumor necrosis factor (TNF) alpha-receptor 1.
Tumor Necrosis Factor Measurement #2 | Week 4
  Measurement of circulating levels of soluble TNF alpha-receptor 2.
Pain Measurement | Week 8
  Pain will be measured with components of the EPHect participant questionnaire using the VAS pain score. Scores range from 0 to 10, higher score is more pain (worse).
Pain Measurement | Week 8
  Pain will be measured with components of the EPHect participant questionnaire using the pain catastrophizing scale. Scores range from 0 to 52, higher scores indicate a greater amount of catastrophizing (worse).
Pain Measurement | Week 8
  Pain will be measured with components of the EPHect participant questionnaire using the mean number of analgesic and/or opioid pills taken per week.
Quality of Life Questionnaire | Week 8
  Physical and mental QOL components will be measured with the Endometriosis Health Profile Questionnaire. Scores range from 0 to 100, higher scores reflect more symptoms and worse health status.
Quality of Life Survey | Week 8
  Physical and mental QOL components will be measured with the Short Form-12 survey. There are two components, a physical component summary (PCS) and a mental health component summary (MCS). Both have a range of 0 to 100, higher scores represent better health.
Inflammatory Markers | Week 8
  Measurement of circulating levels of inflammatory markers (interleukin (IL)-6 and IL-1β.
Protein Measurement | Week 8
  Measurement of circulating levels of high sensitivity-C-reactive protein.
Tumor Necrosis Factor Measurement | Week 8
  Measurement of circulating levels of soluble tumor necrosis factor (TNF) alpha-receptor 1.
Tumor Necrosis Factor Measurement #2 | Week 8
  Measurement of circulating levels of soluble TNF alpha-receptor 2.
Pain Measurement | Week 12
  Pain will be measured with components of the EPHect participant questionnaire using the VAS pain score. Scores range from 0 to 10, higher score is more pain (worse).
Pain Measurement | Week 12
  Pain will be measured with components of the EPHect participant questionnaire using the pain catastrophizing scale. Scores range from 0 to 52, higher scores indicate a greater amount of catastrophizing (worse).
Pain Measurement | Week 12
  Pain will be measured with components of the EPHect participant questionnaire using the mean number of analgesic and/or opioid pills taken per week.
Quality of Life Questionnaire | Week 12
  Physical and mental QOL components will be measured with the Endometriosis Health Profile Questionnaire. Scores range from 0 to 100, higher scores reflect more symptoms and worse health status.
Quality of Life Survey | Week 12
  Physical and mental QOL components will be measured with the Short Form-12 survey. There are two components, a physical component summary (PCS) and a mental health component summary (MCS). Both have a range of 0 to 100, higher scores represent better health.
inflammatory Markers | Week 12
  Measurement of circulating levels of inflammatory markers (interleukin (IL)-6 and IL-1β.
Protein Measurement | Week 12
  Measurement of circulating levels of high sensitivity-C-reactive protein.
Tumor Necrosis Factor Measurement | Week 12
  Measurement of circulating levels of soluble tumor necrosis factor (TNF) alpha-receptor 1.
Tumor Necrosis Factor Measurement #2 | Week 12
  Measurement of circulating levels of soluble TNF alpha-receptor 2.

SECONDARY OUTCOMES:
Pain Measurement | 6 months
  Pain will be measured with components of the EPHect participant questionnaire using the VAS pain score. Scores range from 0 to 10, higher score is more pain (worse).
Pain Measurement | 12 months
  Pain will be measured with components of the EPHect participant questionnaire using the VAS pain score. Scores range from 0 to 10, higher score is more pain (worse).
Qualify of Life Questionnaire | 6 months
  Physical and mental QOL components will be measured with the Endometriosis Health Profile Questionnaire. Scores range from 0 to 100, higher scores reflect more symptoms and worse health status.
Quality of Life Questionnaire | 12 months
  Physical and mental QOL components will be measured with the Endometriosis Health Profile Questionnaire. Scores range from 0 to 100, higher scores reflect more symptoms and worse health status.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Harris, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant information or blood samples could be used for future research studies or sent to other investigators for future research studies without additional consent from participants. These future research studies will be reviewed by an oversight group known as an institutional review board if required by law. The information that identifies participants will first be removed from the information or blood samples. If participants do not want their information or blood samples to be used for future research studies without their consent, interested persons should not participate in this study.
Time Frame: Data will be collected and stored indefinitely.
Access Criteria: Researchers requesting samples in the repository may apply via the completion of a material/data use agreement.